CLINICAL TRIAL: NCT06908863
Title: Cortical Correlations Between Fine Manual Motor Skills and Speech Articulation : Pilot Study
Brief Title: Correlations Between Fine Manual Motor Skills and Speech Articulation
Acronym: MOFiA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24-AOIP-03
Record Dates: First submitted 2025-03-25; First posted 2025-04-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Correlations Between Cerebral Motor Control During a Manual Task and During an Articulatory Task
Keywords: Motor skills, speech, cortical
MeSH Terms: conditions — Speech | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Category 2 pilot study involving healthy subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Motor tasks and oral and facial language (Experimental): Exercises and MRI
  Interventions: Other: Tasks learning and MRI scan

INTERVENTIONS:
Other: Tasks learning and MRI scan — - 2-week learning and training phase of motor tasks and oral and facial language (OLF) tasks.
  Manual fine motor tasks will correspond to activities requiring increasing precision and different types of grip (crushing a ball, modelling clay with the palm of the hand, sorting round coins with thumb/index pliers).
  The OLF praxis tasks will correspond to coordinated movements of different parts of the face (cheeks, lips and tongue).
  - MRI (magnetic resonance imaging) exam, During this exam, the investigator will give to the subject instructions for a task to be carried out. These tasks will correspond to the motor tasks previously trained.

SUMMARY:
The aim of this study is to examine the relationship between cerebral motor control during a manual task and during an articulary task, using functional MRI in a cohort or young adults aged between 18 and 35.

The literature reveals a well-established relationship between manual motor skills and speech from an anatomical and functional point of view. Some studies indicate a proximity between the motor cortical regions corresponding to the hand and the mouth, with a mutual interaction of the two functions from the earliest stages of life (for example, the Babkin reflex). Experimental data shows that hand movements can be influenced by mouth movements. Neurophysiological studies have demonstrated the existence of a link between these two systems in humans and monkeys.

To date, no study has identified the common cortical networks that are active during these two limb movements in a given sample of subjects. The aim of this study is to determine whether such networks exist. The results could be therapeutically relevant, particularly for stroke patients, by enabling more effective restoration of articulatory abilities through complementary limb movements.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18 and 35
2. Right-handed
3. Member of beneficiary of a social security insurance
4. Signature of an informed consent

Exclusion Criteria:

1. Disorders of fine manual motor skills and/or articulatory disorders
2. A neurological history that has affected the subject's cerebral function (stroke, head injury)
3. Contraindication to MRI (presence of ferromagnetic material in the body, claustrophobia)
4. Pregnant women
5. Taking medication that may alter the cerebral haemodynamic signal

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Recording of brain activity during manual motor skills and speech articulation | 2 weeks after inclusion
  Detection and comparison of fMRI image sequences of brain areas based on variations in the difference between oxygenated and deoxygenated hemoglobin during manual motor tasks and silent phoneme articulation

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume SACCO, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, PACA, France

IPD SHARING:
Plan to Share IPD: No